CLINICAL TRIAL: NCT05264168
Title: Prediction of the COBRRA VTE Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-COBRRA-VT
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; DVT
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism | interventions — Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rivaroxaban: Reference group
  Interventions: Drug: Rivaroxaban
- Apixaban: Exposure group
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Rivaroxaban — Any rivaroxaban dispensing claim is used as the reference group
  Other Names: Xarelto
  Groups: Rivaroxaban
Drug: Apixaban — Any apixaban dispensing claim is used as the exposure group
  Other Names: Eliquis
  Groups: Apixaban

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for PE or Proximal DVT [Day -14, Day 0]
* At least 18 years of age

Exclusion Criteria:

* Prior use of a DOAC or warfarin [Day -180, Day 0]
* Stage 4 or 5 chronic kidney disease or end-stage renal disease [Day -180, Day 0]
* Dialysis or renal transplant [Day -180, Day 0]
* Recent major or clinically relevant non-major bleeding [Day -180, Day 0]
* Cancer [Day -180, Day 0]
* Bypass surgery, obesity, or the use of a weight loss or appetite suppressor [Day -180, Day 0]
* Significant liver disease and coagulopathy [Day -180, Day 0]
* Use of CYP3A4 or P-gp inhibitors or inducers [Day -180, Day 0]
* Other indications for anticoagulation (atrial fibrillation or prosthetic heart valve) [Day -180, Day 0]
* Pregnancy or breastfeeding [Day -180, Day 0]
* Use of an antiplatelet [Day -180, Day 0]

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to apixaban users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or apixaban (index date). Analysis is restricted to patients hospitalized with a VTE.
Sampling Method: Non-Probability Sample
Enrollment: 41875 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Relative hazard of major bleeding or clinically relevant non-major bleeding events | Through study completion or censoring, up to 90 days
  Claims-based algorithm: relative hazard of major bleeding or clinically relevant non-major bleeding events

SECONDARY OUTCOMES:
Relative hazard of major bleeding | Through study completion or censoring, up to 90 days
  Claims-based algorithm: relative hazard of major bleeding
Relative hazard of clinically relevant non-major bleeding | Through study completion or censoring, up to 90 days
  Claims-based algorithm: relative hazard of clinically relevant non-major bleeding
Relative hazard of all-cause mortality | Through study completion, up to 90 days
  Claims-based algorithm: relative hazard of all-cause mortality
Relative hazard of recurrent VTE | Through study completion, up to 90 days
  Claims-based algorithm: relative hazard of recurrent VTE
Relative hazard of extracranial bleeding | Through study completion, up to 90 days
  Claims-based algorithm: relative hazard of extracranial bleeding
Relative hazard of intracranial bleeding | Through study completion, up to 90 days
  Claims-based algorithm: relative hazard of intracranial bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT05264168/Prot_SAP_001.pdf